CLINICAL TRIAL: NCT00966823
Title: Phase 2 Fetal Tracheal Balloon (IDE G080077) Study in Diaphragmatic Hernia
Brief Title: Fetal Tracheal Balloon Study in Diaphragmatic Hernia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Device no longer available
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Francois Luks, Francois I. Luks, MD, PhD, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G080077
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Diaphragmatic Hernia; Lung Disease
Keywords: Diaphragm; Trachea; Lung development; Lung growth; Tracheal occlusion; ECMO; Neonatal death
MeSH Terms: conditions — Hernia, Diaphragmatic; Lung Diseases; Tracheal Diseases; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Detachable balloon (Experimental): Intervention: Fetuses treated with endoscopic tracheal occlusion
  Interventions: Device: Fetal tracheal obstruction with detachable balloon (device)

INTERVENTIONS:
Device: Fetal tracheal obstruction with detachable balloon (device) — Fetal tracheal obstruction with detachable balloon (device): Endoscopic placement of a detachable balloon in the fetal trachea at 28-30 weeks gestation.
  - Ultrasound-guided puncture of balloon or, if not feasible, repeat endoscopic tracheoscopy with puncture and retrieval of the balloon at 34 weeks gestation.
  Other Names: Goldvalve Balloon, nFocus Neuromedical, Inc.

SUMMARY:
The purpose of this phase 2 limited study is to examine whether prenatal intervention correct the lung underdevelopment associated with severe diaphragmatic hernia.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) has traditionally been associated with very high mortality rates. Most infants died of pulmonary hypoplasia and severe pulmonary hypertension. This led to correction of CDH and pulmonary hypoplasia before birth. Unfortunately, maternal morbidity of open fetal surgery was significant and fetal mortality was very high (>60%). Moreover, the results of postnatal therapy for CDH improved dramatically, from less than 20% survival several decades ago to more than 70% today.

Fetal intervention has evolved as well, to a minimally invasive approach that involves a single endoscopic port and occlusion of the fetal trachea. While this has considerably decreased the morbidity and fetal mortality of the in utero procedure, its results do not exceed the overall (i.e., non-stratified) results of contemporary postnatal treatment. Most recently, a multicentric cooperative study under (Eurofoetus) has conducted a clinical trial comparing postnatal treatment with endoscopic fetal tracheal occlusion for the most severe forms of CDH. Results of the Eurofoetus trial and of a recent retrospective review involving European and North-American centers have shown the following: 1) It is possible to identify a specific subgroup of fetuses with CDH in whom survival can be predicted to be less than 10%, despite all current methods of postnatal treatment, 2) Survival of fetuses with predicted postnatal survival of 8% was >50% following endoscopic fetal tracheal occlusion, and 3) Fetal tracheal occlusion in that group resulted in an increase in lung size (LHR), from an average of 0.7 pre-intervention, to 1.7 post-intervention.

Based on the available research literature, the results of the Eurofoetus trial, and this institution's experience with endoscopic fetal surgery, we hypothesize that in the highest risk group of fetuses with congenital diaphragmatic hernia, where chances of survival is estimated at less than 10%, endoscopic fetal tracheal occlusion in late second trimester, with reversal of occlusion in mid-third trimester, allows catch-up lung growth and maturation and converts the condition into one with intermediate to good prognosis (predicted survival 50-60%). We propose to offer this form of treatment, under an FDA-approved Investigational Device Exemption (G080077), to eligible patients, on a case-by-case basis, after discussion before a multidisciplinary board.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancies
* Isolated congenital diaphragmatic hernia
* Normal karyotype (amniocentesis)
* Initial diagnosis before 26 weeks gestation
* Competent cervix
* Severity of CDH: lung-to-head ratio (LHR) ≤0.8 at 22-26 weeks gestation
* Liver herniation in the chest
* Informed consent

Exclusion Criteria:

* Preterm labor, premature rupture of membranes or amniotic leak
* Significant maternal morbidity
* Minor (<18 years)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francois I Luks, MD, PhD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital/Women & Infants' Hospital of Rhode Island, Providence, Rhode Island, United States

REFERENCES:
- [Background] Bealer JF, Skarsgard ED, Hedrick MH, Meuli M, VanderWall KJ, Flake AW, Adzick NS, Harrison MR. The 'PLUG' odyssey: adventures in experimental fetal tracheal occlusion. J Pediatr Surg. 1995 Feb;30(2):361-4; discussion 364-5. doi: 10.1016/0022-3468(95)90590-1. PMID 7738765
- [Background] Luks FI, Roggin KK, Wild YK, Piasecki GJ, Rubin LP, Lesieur-Brooks AM, De Paepe ME. Effect of lung fluid composition on type II cellular activity after tracheal occlusion in the fetal lamb. J Pediatr Surg. 2001 Jan;36(1):196-201. doi: 10.1053/jpsu.2001.20051. PMID 11150464
- [Background] Luks FI, Wild YK, Piasecki GJ, De Paepe ME. Short-term tracheal occlusion corrects pulmonary vascular anomalies in the fetal lamb with diaphragmatic hernia. Surgery. 2000 Aug;128(2):266-72. doi: 10.1067/msy.2000.107373. PMID 10923003
- [Background] Wild YK, Piasecki GJ, De Paepe ME, Luks FI. Short-term tracheal occlusion in fetal lambs with diaphragmatic hernia improves lung function, even in the absence of lung growth. J Pediatr Surg. 2000 May;35(5):775-9. doi: 10.1053/jpsu.2000.6067. PMID 10813348
- [Background] De Paepe ME, Johnson BD, Papadakis K, Luks FI. Lung growth response after tracheal occlusion in fetal rabbits is gestational age-dependent. Am J Respir Cell Mol Biol. 1999 Jul;21(1):65-76. doi: 10.1165/ajrcmb.21.1.3511. PMID 10385594
- [Background] De Paepe ME, Papadakis K, Johnson BD, Luks FI. Fate of the type II pneumocyte following tracheal occlusion in utero: a time-course study in fetal sheep. Virchows Arch. 1998 Jan;432(1):7-16. doi: 10.1007/s004280050128. PMID 9463582
- [Background] De Paepe ME, Johnson BD, Papadakis K, Sueishi K, Luks FI. Temporal pattern of accelerated lung growth after tracheal occlusion in the fetal rabbit. Am J Pathol. 1998 Jan;152(1):179-90. PMID 9422535
- [Background] Papadakis K, Luks FI, De Paepe ME, Piasecki GJ, Wesselhoeft CW Jr. Fetal lung growth after tracheal ligation is not solely a pressure phenomenon. J Pediatr Surg. 1997 Feb;32(2):347-51. doi: 10.1016/s0022-3468(97)90208-6. PMID 9044151
- [Background] Luks FI, Deprest JA, Gilchrist BF, Peers KH, van der Wildt B, Steegers EA, Vandenberghe K. Access techniques in endoscopic fetal surgery. Eur J Pediatr Surg. 1997 Jun;7(3):131-4. doi: 10.1055/s-2008-1071072. PMID 9241495
- [Background] Jani JC, Nicolaides KH, Gratacos E, Valencia CM, Done E, Martinez JM, Gucciardo L, Cruz R, Deprest JA. Severe diaphragmatic hernia treated by fetal endoscopic tracheal occlusion. Ultrasound Obstet Gynecol. 2009 Sep;34(3):304-10. doi: 10.1002/uog.6450. PMID 19658113
- [Background] Deprest JA, Flemmer AW, Gratacos E, Nicolaides K. Antenatal prediction of lung volume and in-utero treatment by fetal endoscopic tracheal occlusion in severe isolated congenital diaphragmatic hernia. Semin Fetal Neonatal Med. 2009 Feb;14(1):8-13. doi: 10.1016/j.siny.2008.08.010. Epub 2008 Oct 8. PMID 18845492
- [Background] Yang SH, Nobuhara KK, Keller RL, Ball RH, Goldstein RB, Feldstein VA, Callen PW, Filly RA, Farmer DL, Harrison MR, Lee H. Reliability of the lung-to-head ratio as a predictor of outcome in fetuses with isolated left congenital diaphragmatic hernia at gestation outside 24-26 weeks. Am J Obstet Gynecol. 2007 Jul;197(1):30.e1-7. doi: 10.1016/j.ajog.2007.01.016. PMID 17618746
- [Background] Luks FI, Carr SR, Muratore CS, O'Brien BM, Tracy TF. The pediatric surgeons' contribution to in utero treatment of twin-to-twin transfusion syndrome. Ann Surg. 2009 Sep;250(3):456-62. doi: 10.1097/SLA.0b013e3181b45794. PMID 19644353

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant met inclusion criteria and was enrolled, but was excluded immediately before intervention (active labor), and was therefore excluded from the trial.
Groups:
- Detachable Balloon: Fetuses treated with endoscopic tracheal occlusion
  Fetal tracheal obstruction with detachable balloon (device): - Endoscopic placement of a detachable balloon in the fetal trachea at 28-30 weeks gestation.
  - Ultrasound-guided puncture of balloon or, if not feasible, repeat endoscopic tracheoscopy with puncture and retrieval of the balloon at 34 weeks gestation.
Period: Overall Study
Arm/Group | Detachable Balloon
Started | 3
Completed | 2
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Detachable Balloon
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Newborn Survival at Birth
Time Frame: Newborn period (1 day)
Measure: Number; unit: Participants
Arm/Group | Detachable Balloon
Number analyzed (Participants) | 2
Participants | 1

2. Secondary Outcome: Newborn Survival at 30 Days
Time Frame: 30 days
Population: 1 of 2 enrolled participants (fetuses) survived until birth (Primary outcome). This 1 participant (infant) also survived at 30 days (secondary outcome).
Measure: Number; unit: Participants
Arm/Group | Detachable Balloon
Number analyzed (Participants) | 2
Participants | 1

3. Secondary Outcome: Maternal Complications
Time Frame: Intervention to 30 days postpartum
Measure: Number; unit: occurrences
Arm/Group | Detachable Balloon
Number analyzed (Participants) | 2
occurrences | 0

4. Secondary Outcome: Fetal Morbidity
Description: Fetal morbidity, fetal mortality
Time Frame: Intervention to delivery
Measure: Number; unit: Participants
Arm/Group | Detachable Balloon
Number analyzed (Participants) | 2
Participants | 1

5. Secondary Outcome: Number of Participants With In Utero Lung Growth (LHR) >1.4
Description: Inclusion criterion for the study is LHR<0.9 (extreme pulmonary hypoplasia). Given that LHR is relatively constant during 2nd and 3rd trimester of gestation, "In utero lung growth" is defined as LHR>1.4 (definition of mild/moderate pulmonary hypoplasia) within 2 weeks of intervention.
  Outcome measure = number of participants with LHR>1.4 at 2 weeks post-intervention
Time Frame: Intervention to 2 weeks post-intervention
Measure: Number; unit: Participants
Arm/Group | Detachable Balloon
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: Data collected up to 6 months postnatally
Arm/Group | Detachable Balloon
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes